CLINICAL TRIAL: NCT00617851
Title: A Phase III, Randomized, Controlled, Observer-Blind, Single-Center Study to Evaluate the Consistency of Three Consecutive Lots of a Trivalent Subunit Influenza Vaccine Produced in Embryonated Hen Eggs in Healthy Subjects Aged 18 to 49 Years
Brief Title: Study to Evaluate the Consistency of Three Consecutive Production Lots of Influenza Vaccine in Healthy Subjects 18 to 49 Years Old
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V71P6; 13299
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Results first posted 2010-06-24 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Influenza
Keywords: Influenza; adults; different lots; trivalent subunit influenza virus vaccine (IVV); trivalent subunit influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Influenza virus vaccine (lot A) (Experimental): Lot A of the investigational influenza virus vaccine
  Interventions: Biological: Lot A of Influenza virus vaccine
- Influenza virus vaccine (lot B) (Experimental): Lot B of the investigational influenza virus vaccine
  Interventions: Biological: Lot B of Influenza virus vaccine
- Influenza virus vaccine (lot C) (Experimental): Lot C of the investigational influenza virus vaccine
  Interventions: Biological: Lot C of Influenza virus vaccine
- Influenza virus vaccine (pooled) (Experimental): Pooled data of all three lots (Lot A, B and C) of the investigational influenza virus vaccine
  Interventions: Biological: All 3 consecutive lots of influenza virus vaccine pooled
- Comparator influenza vaccine (Active Comparator): A US licensed influenza virus vaccine
  Interventions: Biological: Comparator influenza virus vaccine

INTERVENTIONS:
Biological: Lot A of Influenza virus vaccine — 1 injection of the trivalent subunit influenza virus vaccine (lot A) administered intramuscularly
  Arms: Influenza virus vaccine (lot A)
Biological: Lot B of Influenza virus vaccine — 1 injection of the trivalent subunit influenza virus vaccine (lot B) administered intramuscularly
  Arms: Influenza virus vaccine (lot B)
Biological: Lot C of Influenza virus vaccine — 1 injection of the trivalent subunit influenza virus vaccine (lot C) administered intramuscularly
  Arms: Influenza virus vaccine (lot C)
Biological: Comparator influenza virus vaccine — 1 injection of the trivalent subunit influenza virus vaccine administered intramuscularly
  Arms: Comparator influenza vaccine
Biological: All 3 consecutive lots of influenza virus vaccine pooled — 1 injection of the pooled trivalent subunit influenza virus vaccine administered intramuscularly
  Arms: Influenza virus vaccine (pooled)

SUMMARY:
The purpose of this research is to demonstrate immunologic equivalence of three consecutive production lots of the subunit influenza vaccine compared to egg-derived inactivated influenza vaccine in healthy subjects 18 to 49 years of ages. In addition, this study is to show how safe and well tolerated a conventional inactivated subunit influenza vaccine, licensed in many countries outside the United States, is compared to an inactivated influenza vaccine, licensed in the United States.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 49 years of age;
* In good health as determined by medical history and physical examination;
* Able and willing to provide written informed consent prior to any study procedure;
* Able to comply with all study procedures and available for all clinic visits scheduled in the study.

Exclusion Criteria:

* Any serious disease, such as: cancer, autoimmune disease (including rheumatoid arthritis), advanced arteriosclerotic disease or complicated diabetes mellitus
* History of any anaphylaxis, serious vaccine reactions, or hypersensitivity to eggs, egg protein, chicken feathers, influenza viral protein, neomycin, polymyxin, or any other vaccine component, chemically related substance, or component of the potential packaging materials (latex);
* Known or suspected impairment/alteration of immune function
* Receipt of an influenza vaccine within 6 months prior to Visit 1;
* Current drug or alcohol abuse or a history of drug or alcohol abuse that in the investigator's opinion would interfere with safety of the subject or the evaluation of the study objectives;
* Laboratory-confirmed influenza disease within 6 months prior to Visit 1

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1507 (Actual)
Dates: Start 2007-11; Primary Completion 2007-12 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Director — Novartis
Locations (2):
- Dominican Republic (2):
  - Centro de Salud Galvan, Santo Domingo
  - Hosp. Nuestra Sra. Altagracia, Santo Domingo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 1 Center along with a satellite center in the Dominican Republic.
Groups:
- Influenza Virus Vaccine (Lot A): One injection of lot A of the investigational influeza virus vaccine
- Influenza Virus Vaccine (Lot B): One injection of lot B of the investigational influeza virus vaccine
- Influenza Virus Vaccine (Lot C): One injection of lot C of the investigational influeza virus vaccine
- Comparator Influenza Vaccine: One injection of the comparator influeza virus vaccine
Period: Overall Study
Arm/Group | Influenza Virus Vaccine (Lot A) | Influenza Virus Vaccine (Lot B) | Influenza Virus Vaccine (Lot C) | Comparator Influenza Vaccine
Started | 430 | 431 | 429 | 217
Completed | 383 | 391 | 384 | 192
Not Completed | 47 | 40 | 45 | 25
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 14 | 7 | 12 | 4
Not completed — Lost to Follow-up | 27 | 29 | 31 | 19
Not completed — Inappropriate Enrollment | 5 | 4 | 1 | 1
Not completed — Unable to classify | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Influenza Virus Vaccine (Lot A): One injection of lot A of the investigational influenza virus vaccine
- Influenza Virus Vaccine (Lot B): One injection of lot B of the investigational influenza virus vaccine
- Influenza Virus Vaccine (Lot C): One injection of lot C of the investigational influenza virus vaccine
- Comparator Influenza Vaccine: One injection of the comparator influenza virus vaccine
- Total: Total of all reporting groups
Arm/Group | Influenza Virus Vaccine (Lot A) | Influenza Virus Vaccine (Lot B) | Influenza Virus Vaccine (Lot C) | Comparator Influenza Vaccine | Total
Number analyzed (Participants) | 430 | 431 | 429 | 217 | 1507
Age Continuous [Mean (Standard Deviation); unit: years] | 31.1 (8.8) | 31.2 (8.6) | 31.3 (8.9) | 31.3 (8.7) | 31.2 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 309 | 306 | 291 | 154 | 1060
  Male | 121 | 125 | 138 | 63 | 447
Race/Ethnicity, Customized [Number; unit: participants]
  Arabic | 1 | 0 | 0 | 0 | 1
  Black | 7 | 11 | 9 | 3 | 30
  Caucasian | 1 | 2 | 1 | 0 | 4
  Hispanic | 421 | 418 | 418 | 214 | 1471
  Native Amer/Alaskan | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs), by Vaccine Lots
Description: The immunologic equivalence of three consecutive production lots of the influenza virus vaccine was measured in terms of GMTs for all vaccine influenza strains.
Time Frame: 21 days after vaccination
Population: The analysis was performed on the per-protocol population, defined as all subjects enrolled who:
  * received all the relevant doses of vaccine correctly, and
  * provided evaluable serum samples at the relevant time points, and
  * had no major protocol deviation
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Influenza Virus Vaccine (Lot A) | Influenza Virus Vaccine (Lot B) | Influenza Virus Vaccine (Lot C)
Number analyzed (Participants) | 393 | 396 | 393
Titers
  Strain A/H1N1 | 566 [503 to 637] | 518 [461 to 582] | 513 [454 to 581]
  Strain A/H3N2 | 352 [318 to 390] | 313 [282 to 348] | 359 [326 to 396]
  Strain B | 99 [89 to 110] | 93 [84 to 104] | 86 [77 to 96]
Statistical Analysis 1: Comparison: Influenza Virus Vaccine (Lot A) vs Influenza Virus Vaccine (Lot B); H01 LotA ≠ LotB versus H1 LotA = LotB H0 refers to the null hypothesis of non-equivalence (inconsistency) in that the two-sided 95% confidence interval (CI) on the geometric mean titer (GMT) ratio is outside the equivalence range (0.67 to 1.5). H1 refers to the alternative hypothesis of equivalence (consistency) in that the two-sided 95% CI on the GMT ratio is within the equivalence range (0.67 to 1.5); Test type: Non-Inferiority or Equivalence — The GMTs and 95% CIs and median, min and max values were calculated for each vaccine group and for each strain by exponentiating (base 10) the least square means of the log transformed (base 10) titers and their 95% CIs obtained from a two-way ANOVA with factors for vaccine group. The overall power is 80.56%, and thus each single test (# of comparisons=9) is performed with a power of 97.62% assuming independency. To account for dropouts, >= 428 subjects per lot was recruited; ANOVA; Ratio of GMTs (A/H1N1 Strain) = 1.09, 95% CI 2-sided [0.92 to 1.29] — The control vaccine arm (Comparator, n=216) is included primarily to provide a comparative assessment for safety rather than for immunogenicity. Sample size calculations were done by means of Nquery Advisor 5.0
Statistical Analysis 2: Comparison: Influenza Virus Vaccine (Lot A) vs Influenza Virus Vaccine (Lot C); H02 LotA ≠ LotC versus H12 LotA = Lotc H0 refers to the null hypothesis of non-equivalence (inconsistency) in that the two-sided 95% CI on the GMT ratio is outside the equivalence range (0.67 to 1.5). H1 refers to the alternative hypothesis of equivalence (consistency) in that the two-sided 95% CI on the GMT ratio is within the equivalence range (0.67 to 1.5); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Ratio of GMTs (A/H1N1 Strain) = 1.1, 95% CI 2-sided [0.93 to 1.31] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Influenza Virus Vaccine (Lot B) vs Influenza Virus Vaccine (Lot C); H03 LotB ≠ LotC versus H13 LotB = LotC H0 refers to the null hypothesis of non-equivalence (inconsistency) in that the two-sided 95% CI on the GMT ratio is outside the equivalence range (0.67 to 1.5). H1 refers to the alternative hypothesis of equivalence (consistency) in that the two-sided 95% CI on the GMT ratio is within the equivalence range (0.67 to 1.5); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Ratio of GMTs (A/H1N1 Strain) = 1.01, 95% CI 2-sided [0.85 to 1.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Influenza Virus Vaccine (Lot A) vs Influenza Virus Vaccine (Lot B); H03 LotA ≠ LotB versus H13 LotA = LotB H0 refers to the null hypothesis of non-equivalence (inconsistency) in that the two-sided 95% CI on the GMT ratio is outside the equivalence range (0.67 to 1.5). H1 refers to the alternative hypothesis of equivalence (consistency) in that the two-sided 95% CI on the GMT ratio is within the equivalence range (0.67 to 1.5); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Ratio of GMTs (A/H3N2 Strain) = 1.12, 95% CI 2-sided [0.97 to 1.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Influenza Virus Vaccine (Lot A) vs Influenza Virus Vaccine (Lot C); H03 LotA ≠ LotC versus H13 LotA = LotC H0 refers to the null hypothesis of non-equivalence (inconsistency) in that the two-sided 95% CI on the GMT ratio is outside the equivalence range (0.67 to 1.5). H1 refers to the alternative hypothesis of equivalence (consistency) in that the two-sided 95% CI on the GMT ratio is within the equivalence range (0.67 to 1.5); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Ratio of GMTs (A/H3N2 strain) = 0.98, 95% CI 2-sided [0.85 to 1.13] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Influenza Virus Vaccine (Lot B) vs Influenza Virus Vaccine (Lot C); [analysis description as in outcome 1, analysis 3]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Ratio of GMTs (A/H3N2 strain) = 0.87, 95% CI 2-sided [0.76 to 1.01] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Influenza Virus Vaccine (Lot A) vs Influenza Virus Vaccine (Lot B); [analysis description as in outcome 1, analysis 4]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Ratio of GMTs (B strain) = 1.06, 95% CI 2-sided [0.91 to 1.23] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Influenza Virus Vaccine (Lot A) vs Influenza Virus Vaccine (Lot C); [analysis description as in outcome 1, analysis 5]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Ratio of GMTs (B strain) = 1.15, 95% CI 2-sided [0.99 to 1.33] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Influenza Virus Vaccine (Lot B) vs Influenza Virus Vaccine (Lot C); [analysis description as in outcome 1, analysis 3]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Ratio of GMTs (B strain) = 1.09, 95% CI 2-sided [0.94 to 1.26] — The control vaccine arm (n=216) is included primarily to provide a comparative assessment for safety rather than for immunogenicity. Sample size calculations were done by means of Nquery Advisor 5.0

2. Secondary Outcome: Geometric Mean Titers (GMTs), by Vaccine Group and Strain
Description: The GMTs and 95% CIs were calculated for each of the vaccine group (three consecutive production lots pooled for the investigational influenza virus vaccine and comparator) and for each strain.
Time Frame: 21 days after vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- Influenza Virus Vaccine (Strain A/H1N1): One injection of the investigational influenza virus vaccine-Strain A/H1N1
- Influenza Virus Vaccine (Strain A/H3N2): One injection of the investigational influenza virus vaccine-Strain A/H3N2
- Influenza Virus Vaccine (Strain B): One injection of the investigational influenza virus vaccine-Strain B
- Comparator Influenza Vaccine (Strain A/H1N1): One injection of the comparator influenza virus vaccine-Strain A/H1N1
- Comparator Influenza Vaccine (Strain A/H3N2): One injection of the comparator influenza virus vaccine-Strain A/H3N2
- Comparator Influenza Vaccine (Strain B): One injection of the comparator influenza virus vaccine-Strain B
Arm/Group | Influenza Virus Vaccine (Strain A/H1N1) | Influenza Virus Vaccine (Strain A/H3N2) | Influenza Virus Vaccine (Strain B) | Comparator Influenza Vaccine (Strain A/H1N1) | Comparator Influenza Vaccine (Strain A/H3N2) | Comparator Influenza Vaccine (Strain B)
Number analyzed (Participants) | 1182 | 1182 | 1182 | 194 | 194 | 194
titers | 532 [497 to 570] | 341 [321 to 361] | 93 [87 to 98] | 799 [666 to 957] | 683 [590 to 790] | 99 [85 to 115]

3. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Symptoms
Description: Solicited local and systemic reactions were assessed after vaccination for the two vaccines (three consecutive production lots pooled for the investigational influenza virus vaccine and comparator) and for each of the three consecutive production lots of the investigational influenza virus vaccine.
Time Frame: 7 days after vaccination
Population: The analysis was performed on the safety population, defined as all subjects who provided post-baseline safety data.
Measure: Number; unit: Participants
Groups:
- Influenza Virus Vaccine (Pooled): One injection of the investigational influenza virus vaccine (all lots pooled)
Arm/Group | Influenza Virus Vaccine (Lot A) | Influenza Virus Vaccine (Lot B) | Influenza Virus Vaccine (Lot C) | Influenza Virus Vaccine (Pooled) | Comparator Influenza Vaccine
Number analyzed (Participants) | 403 | 404 | 402 | 1209 | 202
Participants
  Any Local Reaction | 114 | 96 | 100 | 310 | 54
  Erythema (mm) | 15 | 12 | 17 | 44 | 9
  Induration (mm) | 19 | 19 | 24 | 62 | 12
  Swelling (mm) | 15 | 24 | 14 | 53 | 14
  Ecchymosis (mm) | 14 | 13 | 14 | 41 | 9
  Pain | 96 | 87 | 85 | 268 | 44
  Any Systemic Reaction | 148 | 148 | 147 | 443 | 76
  Chills | 30 | 28 | 29 | 87 | 17
  Malaise | 45 | 52 | 47 | 144 | 25
  Myalgia | 73 | 75 | 65 | 213 | 40
  Arthralgia | 19 | 25 | 25 | 69 | 14
  Headache | 100 | 94 | 98 | 292 | 48
  Sweating | 14 | 14 | 20 | 48 | 9
  Fatigue | 29 | 41 | 41 | 111 | 16
  Fever (≥38C) | 17 | 24 | 13 | 54 | 7

4. Secondary Outcome: Number of Subjects With at Least One Unsolicited Adverse Event
Description: Number of subjects reporting at least one unsolicited adverse event, regardless of the assessement of relatedness to the study vaccines (each of the three consecutive production lots of the investigational influenza virus vaccine, the pooled influenza virus vaccine, and the comparator influenza vaccine).
Time Frame: 3 weeks after vaccination
Population: The analysis was performed on the safety population, defined as all subjects who provided post-baseline safety data.
Measure: Number; unit: participants
Arm/Group | Influenza Virus Vaccine (Pooled) | Comparator Influenza Vaccine | Influenza Virus Vaccine (Lot A) | Influenza Virus Vaccine (Lot B) | Influenza Virus Vaccine (Lot C)
Number analyzed (Participants) | 1209 | 202 | 403 | 404 | 402
participants | 189 | 33 | 56 | 68 | 65

5. Secondary Outcome: Percentage of Subjects With Seroprotection and Seroconversion (Strain A/H1N1)
Description: The percentage of subjects who were seroprotected and seroconverted were considered statistically compliant with the stated CBER guidance criteria if:
  * the lower bound of the two-sided 95% CI for the percentage of seroprotected subjects (HI antibody titer ≥1:40) met or exceeded 70%.
  * the lower bound of the two-sided 95% CI for the percentage of subjects achieving seroconversion rate (prevaccination HI<10/ postvaccination HI ≥40 or at least a fourfold increase in titer from non-negative prevaccination serum [HI≥10]), for HI antibody met or exceeded 40%.
Time Frame: 21 days after vaccination
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentages of participants
Arm/Group | Influenza Virus Vaccine (Lot A) | Influenza Virus Vaccine (Lot B) | Influenza Virus Vaccine (Lot C) | Influenza Virus Vaccine (Pooled) | Comparator Influenza Vaccine
Number analyzed (Participants) | 393 | 396 | 393 | 1182 | 194
percentages of participants
  Seroprotection (HI titer => 40) | 98 [96 to 99] | 99 [97 to 100] | 98 [96 to 99] | 98 [97 to 99] | 98 [95 to 99]
  Seroconversion | 95 [92 to 97] | 94 [92 to 96] | 93 [90 to 95] | 94 [93 to 95] | 96 [92 to 98]

6. Secondary Outcome: Percentage of Subjects With Seroprotection and Seroconversion (Strain A/H3N2)
Description: as for outcome 5
Time Frame: 21 days after vaccination
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentages of participants
Arm/Group | Influenza Virus Vaccine (Lot A) | Influenza Virus Vaccine (Lot B) | Influenza Virus Vaccine (Lot C) | Influenza Virus Vaccine (Pooled) | Comparator Influenza Vaccine
Number analyzed (Participants) | 393 | 396 | 393 | 1182 | 194
percentages of participants
  Seroprotection (HI titer ≥40) | 99 [98 to 100] | 98 [97 to 99] | 99 [98 to 100] | 99 [98 to 100] | 99 [97 to 100]
  Seroconversion | 70 [65 to 74] | 64 [59 to 69] | 68 [63 to 72] | 67 [65 to 70] | 84 [78 to 88]

7. Secondary Outcome: Percentage of Subjects With Seroprotection and Seroconversion (Strain B)
Description: as for outcome 5
Time Frame: 21 days after vaccination
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentages of participants
Arm/Group | Influenza Virus Vaccine (Lot A) | Influenza Virus Vaccine (Lot B) | Influenza Virus Vaccine (Lot C) | Influenza Virus Vaccine (Pooled) | Comparator Influenza Vaccine
Number analyzed (Participants) | 393 | 396 | 393 | 1182 | 194
percentages of participants
  Seroprotection (HI titer ≥40) | 88 [85 to 91] | 88 [85 to 91] | 84 [80 to 87] | 87 [85 to 89] | 90 [85 to 94]
  Seroconversion | 85 [81 to 88] | 86 [82 to 89] | 81 [76 to 84] | 84 [82 to 86] | 86 [80 to 90]

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected for 6 months after vaccination. All adverse events were collected for 21 days after vaccination.
Description: Of the 1507 subjects enrolled and randomized in this study, 96 were not included in the safety analysis (82 in the pooled influenza virus vaccine group and 14 in the comparator influenza vaccine group) as they had no safety data. These subjects have been excluded from the safety analysis to avoid underestimating the incidence rates of reactions.
Arm/Group | Influenza Virus Vaccine (Pooled) | Comparator Influenza Vaccine
Serious Adverse Events (participants affected / at risk) | 11/1209 | 4/202
Other Adverse Events (participants affected / at risk) | 0/1209 | 0/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Influenza Virus Vaccine (Pooled) (N=1209) | Comparator Influenza Vaccine (N=202)
Abortion Induced (Surgical and medical procedures) | 2 (2) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1)
Abscess Limb (Infections and infestations) | 0 (0) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Fibroadenoma of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fractured Coccyx (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gas Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Intracranial Aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Multi-Organ Failure (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less